CLINICAL TRIAL: NCT02481713
Title: Enhancing Adherence to Cognitive Rehabilitation
Brief Title: Improving Adherence to Cognitive Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1790-R
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Psychosis
Keywords: psychosis; adherence; motivation
MeSH Terms: conditions — Psychotic Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MI condition (Experimental): motivational interview condition
  Interventions: Behavioral: motivational interviewing
- CI condition (Sham Comparator): learning style interview condition
  Interventions: Behavioral: learning style interviews

INTERVENTIONS:
Behavioral: motivational interviewing — motivational interviewing
  Arms: MI condition
Behavioral: learning style interviews — interview and feedback about learning style
  Arms: CI condition

SUMMARY:
Purpose of study is to evaluate impact of brief motivational interviewing vs. feedback on learning styles in improving attendance to cognitive training

DETAILED DESCRIPTION:
This study is evaluating whether motivational enhancement can improve outcomes of cognitive rehabilitation in Veterans with schizophrenia spectrum disorders. Approximately 120 individuals will be randomized to either a 2-session motivational interview (MI, experimental condition) or a 2-session assessment and feedback on learning styles (CI, active control), and will then be asked to participate in 4 months of cognitive rehabilitation. Booster MI or CI sessions will be administered monthly over the course of the cognitive rehabilitation. Primary outcome is number of cognitive rehabilitation sessions attended.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of psychotic disorder
* 18 years old or older

Exclusion Criteria:

* meeting criteria for substance abuse/dependence in past 30 days
* psychiatric hospitalization in past 30 days
* change in psychiatric medications in past 30 days
* severe auditory/visual impairment
* evidence of developmental disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M. Fiszdon, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available once primary and secondary study aims have been published.
Access Criteria: Completely de-identified data will be made available to other investigators, with written request and IRB approval, ideally under a data use agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MI Condition | CI Condition
Started | 56 | 58
Completed | 40 | 42
Not Completed | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MI Condition | CI Condition | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.52 (10.40) | 53.34 (12.74) | 55.41 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 43 | 48 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 53 | 53 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 29 | 58
  White | 24 | 26 | 50
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 1 | 0 | 1
Education [Mean (Standard Deviation); unit: years] | 12.52 (2.42) | 13.04 (2.21) | 12.79 (2.32)
Marital status [Count of Participants; unit: Participants]
  ever married | 31 | 29 | 60
  never married | 25 | 29 | 54
Number of hospitalizations [Median (Inter-Quartile Range); unit: hospitalizations] | 4.0 [1.0 to 10.0] | 4.0 [2.0 to 7.0] | 4.0 [1.0 to 10.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Sessions Attended
Description: number of cognitive training sessions attended
Time Frame: end of four month training period
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | MI Condition | CI Condition
Number analyzed (Participants) | 56 | 58
sessions | 7.70 (10.82) | 4.98 (6.63)
Statistical Analysis 1: Comparison: CI Condition; Test type: Non-Inferiority — All analyses were two-tailed with alpha set at 0.05; p = 0.24, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Sessions Attended
Description: number of sessions attended among patients who attended at least 1 session
Time Frame: end of 4 month training period
Population: participants who attended at least 1 cognitive training session
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | MI Condition | CI Condition
Number analyzed (Participants) | 41 | 40
sessions | 10.51 (11.43) | 7.23 (6.91)
Statistical Analysis 1: Comparison: CI Condition; Test type: Superiority; p = .0001, Regression, zero-inflated Poisson; Risk Ratio (RR) = 1.46, 95% CI 2-sided [1.25 to 1.69]

ADVERSE EVENTS:
Time Frame: baseline to end of study participation, approximately 5 months later
Arm/Group | MI Condition | CI Condition
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 4/56 | 4/58
Other Adverse Events (participants affected / at risk) | 1/56 | 1/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MI Condition (N=56) | CI Condition (N=58)
admit/chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
admit/suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
admit/dental (General disorders) | 1 (1) | 0 (0)
admit/abnrml blood (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
admit/sub abuse (Psychiatric disorders) | 1 (1) | 0 (0)
admit/cellulitis (General disorders) | 0 (0) | 1 (1)
admit/lower extr pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
admit/hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MI Condition (N=56) | CI Condition (N=58)
ER/fall (General disorders) | 1 (1) | 0 (0)
ER/suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02481713/Prot_SAP_000.pdf